CLINICAL TRIAL: NCT02683421
Title: Evaluation of Subcutaneous (SC) Injected Tc 99m Tilmanocept Localization in Active Rheumatoid Arthritis (RA) Subjects by SPECT and SPECT/CT Imaging
Brief Title: Evaluation of SC Injected Tc 99m Tilmanocept Localization in Active RA Subjects by SPECT and SPECT/CT Imaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-23
Record Dates: First submitted 2016-01-22; First posted 2016-02-17 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Tilmanocept; Imaging
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Other): Healthy Volunteers: 50 mcg tilmanocept with 2 millicuries (mCi) Tc 99m
  Interventions: Drug: Tilmanocept
- Cohort 2 (Other): Healthy Volunteers: 200 mcg tilmanocept with 2 mCi Tc 99m
  Interventions: Drug: Tilmanocept
- Cohort 3 (Experimental): RA Group: 50 mcg tilmanocept with 2 mCi Tc 99m
  Interventions: Drug: Tilmanocept
- Cohort 4 (Experimental): RA group:200 mcg tilmanocept with 2 mCi Tc 99m
  Interventions: Drug: Tilmanocept

INTERVENTIONS:
Drug: Tilmanocept
  Other Names: Lymphoseek

SUMMARY:
Determine the localization of Tc 99m tilmanocept by SPECT and SPECT/CT imaging in subjects with active RA and concordance with clinical symptomology.

DETAILED DESCRIPTION:
While many types of cells, including T-cells, B-cells, dendritic cells and activated synovial fibroblasts contribute significantly to the establishment and maintenance of the pathology of rheumatoid arthritis (RA), (Ma et al., Noack et al., Bugatti et al., Boissier et al., Tran et al.) macrophages play a critical role in RA (Kinne et al.). They produce most of the tumor necrosis factor alpha (TNFα) that drives and perpetuates the inflammatory cycle in RA (Leizer et al., Westra et al., Hamilton et al., Keffer et al., Noack et al., Bugatti et al., Boissier et al., Tran et al., Kinne et al., Zwerina et al., Feldman et al., Schett et al.). In the synovial sublining of a joint affected by RA, macrophages are the dominant cell type (Kraan et al., Cutolo et al.). In the inflamed joint as a whole, macrophages in RA patients make up at least 30%-40% of all cells (Kennedy et al.). Furthermore, macrophages participate directly in the destruction of bone and cartilage (Ma et al.). Activated macrophage populations and synoviocytes are the predominant cell types at the interface between pannus and cartilage and secrete destructive proteases in abundance (Bresnihan et al.). As a result, it may not be surprising that synovial macrophage numbers-but not the numbers of other immune cell types-correlate with radiographically determined joint destruction in RA (Mulherin et al., Yanni et al.). While macrophages may play a role in other pathologies that cause joint pain and inflammation, the degree to which macrophages are involved in the pathological process of RA and the sheer mass or volume of macrophages that infiltrate the joints inflamed due to RA differentiates RA from other rheumatic diseases. Therefore, detection of the density or numbers of macrophages in inflamed joints may permit differentiation of patients with RA from those with other causes of arthritis. In addition, it is known that the RA pathology begins significantly before, perhaps years before, the onset of symptoms (i.e., joint pain and inflammation) and well before the beginning of bone destruction (Deane et al., El-Gabalawy et al.). Macrophage infiltration of synovial tissues precedes development of clinical signs of RA in animal studies (Kraan et al.). In humans, macrophage infiltrations of synovial tissues are present when RA patients first develop clinical symptoms (Demoruelle et al., van de Sande et al.). Therefore, detection of the density or numbers of macrophages in inflamed joints may facilitate more sensitive and specific identification of RA patients as soon as they present with symptoms and early in the course of their illnesses when DMARDs are likely to be most effective.

An interesting and important observation that has been made in many studies is that the number of macrophages in synovial tissue, and particularly in the synovial sublining, declines in RA patients when they are given DMARD therapy (Hamilton et al.). Furthermore, the degree to which synovial macrophage numbers decline is correlated with the magnitude of the DMARD (DAS28) with changes in sublining macrophage numbers as determined by biopsies and found a significant correlation between the change in the number of macrophages and the change in DAS28 (Pearson correlation 0.874, p < 0.01) ( Haringman et al.). The authors of this study have confirmed these findings in two additional studies, which used slightly different methodologies (Bresnihan et al., Bresnihan et al.). This correlation between declining macrophage numbers and the efficacy of DMARD therapy appears to be largely independent of the kind of DMARD therapy being investigated (Hamilton et al., Kinne et al., Franz et al., Kraan et al., Catrina et al., Cunnane et al., Vieira-Sousa et al.). These findings indicate that assaying the number of macrophages in inflamed joints of patients with RA could be used as an objective measure of the efficacy of DMARD therapy. These findings further suggest that assaying the number of macrophages in inflamed joints of patients with RA could be used in clinical studies as a biomarker of clinical response for potential new RA therapeutics. The problem with current methodologies is that macrophage numbers and densities need to be determined with synovial biopsies. This is obviously an invasive procedure that samples only a small portion of the inflamed synovial tissue and is painful and unpleasant for the patient. What would be preferable and likely more accurate is an imaging protocol, such as the one proposed in this application, that can assay synovial macrophages more completely and less invasively.

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided written informed consent with HIPPA authorization before the initiation of any study-related procedures.

CONTROLS:

* The subject is between 21-45 years of age at the time of consent.
* The subject has not experienced joint pain for at least 4 weeks prior to the consent date and is deemed to be clinically free of any inflammatory disease(s).

ACTIVE RHEUMATOID ARTHRITIS

* The subject is at least 21 years of age at the time of consent.
* The subject has moderate to severe RA, based on either the 1987American College of Rheumatology (ACR) score of ≥ 4/7 or the 2010 ACR/EULAR score of ≥ 6/10.
* The subject has a DAS28 of >4.4 (using the ESR).
* If the subject is on methotrexate, they have been at a stable dose for > 4 weeks prior to the screening visit.
* If the subject is on biologic therapy, they have been at a stable dose > 8 weeks prior to the screening visit.
* If the subject is on non-steroidal anti-inflammatories (NASIDS) or oral corticosteroids, it is ≤ 10mgmg/day or equivalent, and has been at a stable dose for > 4 weeks prior to the screening visit.

Exclusion Criteria:

* The subject is pregnant or lactating.
* BMI >32.0.
* The subject has had or is currently receiving chemotherapy for a non-inflammatory related condition or radiation therapy.

Chronic or persistent infection or has any condition that would, in the opinion of the examining physician, preclude their participation.

* The subject has a known allergy to or has had a reaction to dextran exposure.
* The subject has received an investigational product within 30 days prior to he Tc99m tilmanocept administration.
* The subject has received any radiopharmaceutical within 7 radioactive half-lives of that radiopharmaceutical prior to the administration of Tc 99m tilmanocept.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Principal Investigator — Navidea Biopharmaceuticals
Locations (2):
- United States (2):
  - Axis Clinical Trials, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Subjects: 50 mcg/2 mCi Dose: Healthy Volunteers: 50 mcg tilmanocept with 2 millicuries (mCi) Tc 99m
  Tilmanocept
- Controls Subjects: 200 mcg/2mCi Dose: Healthy Volunteers: 200 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- RA Subjects: 50 mcg/2 mCi Dose: Rheumatoid arthritis (RA) Group: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- RA Subjects: 200 mcg/2 mCi Dose: RA group:200 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
Period: Overall Study
Arm/Group | Control Subjects: 50 mcg/2 mCi Dose | Controls Subjects: 200 mcg/2mCi Dose | RA Subjects: 50 mcg/2 mCi Dose | RA Subjects: 200 mcg/2 mCi Dose
Started | 5 | 4 | 4 | 5
Completed | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Subjects: 50 mcg/20 mCi Dose: Healthy Volunteers: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- Control Subjects: 200 mcg/2 mCi Dose: Healthy Volunteers: 200 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- RA Subjects: 50 mcg/2 mCi Dose: RA Group: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- Total: Total of all reporting groups
Arm/Group | Control Subjects: 50 mcg/20 mCi Dose | Control Subjects: 200 mcg/2 mCi Dose | RA Subjects: 50 mcg/2 mCi Dose | RA Subjects: 200 mcg/2 mCi Dose | Total
Number analyzed (Participants) | 5 | 4 | 4 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 4 | 17
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (7.86) | 32.3 (5.74) | 47 (16.33) | 56.8 (18.54) | 43.2 (15.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 4 | 11
  Male | 4 | 2 | 0 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 4 | 11
  Not Hispanic or Latino | 3 | 3 | 0 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 0 | 5
  White | 2 | 1 | 4 | 4 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 4 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Localization of Tc 99m Tilmanocept by Planar and SPECT/CT Imaging in Subjects With Active RA and Concordance With Swollen/Tender Joints
Description: The primary endpoint was to compare the cumulative total of anatomical zones of active RA (which were clinically defined by a swollen/tender classification during the DAS28 joint count assessment performed at baseline) with Tc 99m tilmanocept localization observed at 2-3 hours and at 4-6 hours after administration on Day 1. Tc 99m tilmanocept localization is defined by accumulation of radioactivity at an intensity greater than background, which was qualitatively determined by the central reader's visual assessment of the acquired images .
Time Frame: Swollen/tender joints assessment at baseline and Tc 99m tilmanocept localization at 2-3 hours and 4-6 hours after administration on Day 1
Measure: Number; unit: Joints
Groups:
- Control Subjects: 50 mcg/2 mCi Dose: Healthy Volunteers: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
Arm/Group | Control Subjects: 50 mcg/2 mCi Dose | Control Subjects: 200 mcg/2 mCi Dose | RA Subjects: 50 mcg/2 mCi Dose | RA Subjects: 200 mcg/2 mCi Dose
Number analyzed (Participants) | 5 | 4 | 4 | 5
Joints
  Total swollen/tender regions at baseline | 0 | 0 | 30 | 35
  Total Tc localized regions at 2-3 hours | 0 | 0 | 1 | 9
  Total Tc localized regions at 4-6 hours | 0 | 0 | 2 | 7

2. Secondary Outcome: Dose-dependent Tc 99m Tilmanocept Localization Intensity by Planar and SPECT/CT Imaging
Description: Tc 99m tilmanocept localization intensity on planar imaging was compared among dose/disease groups. Localization intensity was quantitatively analyzed by observing average voxel intensity in regions of interest, which were drawn over areas of increased uptake in the RA-affected joints.
Time Frame: 2-4 hours and 4-6 hours
Measure: Mean (Standard Deviation); unit: Voxel Intensity
Arm/Group | Control Subjects: 50 mcg/2 mCi Dose | Control Subjects: 200 mcg/2 mCi Dose | RA Subjects: 50 mcg/2 mCi Dose | RA Subjects: 200 mcg/2 mCi Dose
Number analyzed (Participants) | 5 | 4 | 4 | 5
Voxel Intensity
  2-4 Hours | 0.96 (0.483) | 0.97 (0.685) | 1.17 (0.520) | 1.16 (0.694)
  4-6 Hours | 0.97 (0.442) | 1.00 (0.742) | 1.21 (0.422) | 1.13 (0.648)

3. Secondary Outcome: Localization Intensity of Tc 99m Tilmanocept by Planar Imaging in Regions of Interest Relative to Background in All Dose Groups
Description: Tc 99m tilmanocept localization intensity on planar imaging relative to localization intensity in corresponding background regions was calculated (percent of background) for each region of interest and averaged for each dose/disease group.
Time Frame: 2-4 hours and 4-6 hours
Measure: Mean (Standard Deviation); unit: Percent difference from background
Arm/Group | Control Subjects: 50 mcg/2 mCi Dose | Control Subjects: 200 mcg/2 mCi Dose | RA Subjects: 50 mcg/2 mCi Dose | RA Subjects: 200 mcg/2 mCi Dose
Number analyzed (Participants) | 5 | 4 | 4 | 5
Percent difference from background
  2-3 hours | -2.47 (4.471) | -9.21 (5.178) | 1.59 (6.309) | 9.11 (25.939)
  4-6 hours | -1.32 (4.692) | -6.74 (5.326) | 3.31 (14.544) | 16.34 (25.453)

ADVERSE EVENTS:
Groups:
- Cohort 1: Healthy Volunteers: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- Cohort 2: Healthy Volunteers: 200 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- Cohort 3: RA Group: 50 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
- Cohort 4: RA group:200 mcg tilmanocept with 2 mCi Tc 99m
  Tilmanocept
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 1/4 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=4) | Cohort 3 (N=4) | Cohort 4 (N=5)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pain at injection site for 5 days following injection
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — probably related to tilmanocept injection
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — probably related to tilmanocept injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and make modifications to the publication.